CLINICAL TRIAL: NCT03268993
Title: A Phase 0 Study Evaluating the Systemic Bioavailability and Pharmacodynamic Effects of Avmacol® in the Oral Mucosa of Patients Following Curative Treatment for Tobacco-related Head and Neck Cancer
Brief Title: Effects of Avmacol® in the Oral Mucosa of Patients Following Curative Treatment for Tobacco-related Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Arizona (Other)
Responsible Party: Principal Investigator, Dan Zandberg, Principal Investigator, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 18-028
Record Dates: First submitted 2017-07-10; First posted 2017-08-31 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Head and Neck Cancer; Head and Neck Squamous Cell Carcinoma (HNSCC); Head and Neck Carcinoma; Head and Neck; Tobacco-Related Carcinoma; Carcinoma in Situ; Dysplasia; Hyperplasia; Premalignant Lesion
Keywords: prevention; dietary supplement; broccoli; avmacol
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Carcinoma in Situ; Hyperplasia

STUDY DESIGN:
Intervention Model Description: Thirty-six individuals who have previously been treated for tobacco-related, HPV-negative HNSCC will be recruited for this study.
  After being deemed eligible, subjects will be assigned a patient number and be registered into the CTMA database.
  At registration, they will be randomized to receive either 4 tablets/day in Cycle 1 or 8 tablets/day in Cycle 1 (and the other dose in Cycle 2). This randomization is not blinded. Randomization will be stratified by history of head and neck radiation therapy (yes or no).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Avmacol (Other): You will be given a higher dose of Avmacol® each month, taking 2 Avmacol® tablets per day the first month (Cycle 1), 4 Avmacol® tablets per day the second month (Cycle 2), and 8 Avmacol® tablets per day the third month (Cycle 3). Investigators will study how Avmacol® affects your body by collecting three different tissues: 1) your cheek cells (buccal cells); 2) your urine; and 3) your blood. After you have finished three months of Avmacol®, you will return one month later for an end-of-study visit.
  Interventions: Dietary Supplement: Avmacol

INTERVENTIONS:
Dietary Supplement: Avmacol — Avmacol is a dietary supplement available over the counter
  Other Names: broccoli see extract

SUMMARY:
Avmacol is an over-the-counter dietary supplement containing broccoli seed and sprout extracts in tablet form, hypothesized to activate protective cellular pathways including detoxication. In this study, participants who have been curatively treatment for head and neck cancer, will take Avmacol twice a day for 3 months.

DETAILED DESCRIPTION:
The broccoli seed preparation, Avmacol®, results in acute and/or sustained induction of NRF2 target gene transcripts in the oral mucosa of patients who have been curatively treated for a tobacco-related head and neck squamous cell carcinoma (HNSCC), including high grade dysplasia, carcinoma in situ, or invasive carcinoma. This study is not designed to examine the therapeutic or reparative effects of Avmacol® on premalignant lesions of the oral cavity.

We will systematically assess the clinical chemopreventive potential of Avmacol® administration to patients with tobacco-related HNSCC at high risk for second primary tumor by:

1. Conducting this phase 0 clinical study to evaluate the pharmacodynamic range of NRF2 pathway activation in the oral mucosa of HNSCC patients, in response to two tolerable and bioactive doses of Avmacol®;
2. Determining whether the level of NRF2 pathway activation achieved in human oral epithelium is chemopreventive in the NQO1 murine model of environmental carcinogenesis; and
3. Analyzing specimens from the Phase 0 trial to determine whether Avmacol® induces changes in alternative biomarkers of SF chemopreventive efficacy identified in the laboratory.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have completed curative-intent therapy (including surgery, radiation, and/or chemotherapy) for a first tobacco-related oral premalignant lesion (OPL) or HNSCC of any stage (eligible lesions include high grade dysplasia; carcinoma in situ; or stage I-IVa HNSCC).
2. Primary site may include oral cavity, pharynx, or larynx. Oropharynx primaries must be HPV (-) as defined by routine p16 IHC at the local site.
3. Participants may be enrolled between 3 months and 5 years AFTER completion of curative-intent therapy (including surgery, radiotherapy, and/or chemotherapy).
4. Participants may have untreated OPLs (i.e., hyperplasia, dysplasia, carcinoma in situ) at the time of study entry, provided the index OPL or HNSCC was definitively treated.
5. Participants must be at least 18 years old.
6. Participants must have a Karnofsky Performance Status of 80% or higher or an ECOG of 0-1 (Appendix A).
7. Current and former tobacco users are eligible. The tobacco use assessment form must be completed following consent, to assure eligibility (Appendix B). Patients must have ≥10 pack-year cumulative tobacco exposure or its equivalent to be eligible. This is defined as follows:

   1. Cigarette exposure: ≥10 pack-years OR
   2. Cigar exposure: ≥ 10 cigar-years, where 1 cigar year is defined as having smoked on average ≥ 1 cigar/day for a year OR
   3. Chewing tobacco: ≥10 snuff-years, where 1 snuff year is defined as using on average ≥ 1 pinch (dip) of chewing tobacco/day for a year.
8. Able to perform written, informed consent.
9. Women of childbearing potential (WCBP) must have a negative urine pregnancy test within 7 Days prior to the first study intervention.
10. WCBP and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study and for the duration of study participation.

Exclusion Criteria:

1. Participants have a history of another malignancy within 2 years prior to starting study treatment, except for excised and cured carcinoma-in-situ of breast or cervix; non-melanomatous skin cancer; T1-2, N0, M0 differentiated thyroid carcinoma either resected or under active surveillance; superficial bladder cancer; T1a or T1b prostate cancer comprising < 5% of resected tissue with normal prostate specific antigen (PSA) since resection, or status post external beam radiation or brachytherapy with normal PSA since radiation.
2. Primary oropharyngeal HNSCC which is HPV (+) as defined by p16 IHC.
3. Participants with acute intercurrent illness or those who had major surgery within the preceding 4 weeks unless they have fully recovered.
4. Participants who have a positive pregnancy test, are pregnant, or breast feeding.
5. Patients who are not practicing adequate contraception are ineligible if they are of child bearing potential.
6. Patients currently using anti-neoplastic or anti-tumor agents, including chemotherapy, radiation therapy, immunotherapy, and hormonal anticancer therapy.
7. Chronic anticoagulation with warfarin. Patients on low molecular weight heparin or fondaparinux may be enrolled.
8. Use of chronic prescribed medications which are potent inducers or inhibitors of CYP3A4 (Appendix C).
9. Chronic use of steroids at immunosuppressive doses. (Note, physiologic replacement doses of glucocorticoid or mineralocorticoid are acceptable, eg. prednisone 5-10 mg/day; fludrocortisone 0.1-0.2 mg/day.)
10. History of severe food intolerance to broccoli.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-07-27 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2019-07-22 (Actual)

PRIMARY OUTCOMES:
Change in NRF2 target gene expression | From baseline throughout treatment period, up to 4 months
  Quantitative changes in NRF2 target gene transcripts expression (i.e. NQO1 and GCLC) in oral mucosa (buccal cytobrush) by quantitative polymerase chain reaction (qPCR) according to a linear mixed model framework.

SECONDARY OUTCOMES:
Change in NRF2 target proteins | From baseline throughout treatment period, up to 4 months
  Changes in NRF2 target proteins in buccal punch biopsies by immunoblotting.
Change in NRF2 target gene transcripts | From baseline throughout treatment period, up to 4 months
  Change in NRF2 target gene transcripts, between the two doses of Avmacol® by immunoblotting.
Change in NRF2-independent proteins | From baseline throughout treatment period, up to 4 months
  Change in NRF2 target gene transcripts, between the two doses of Avmacol® by immunoblotting.
Alterations of Avmacol® activity in PBMCs - NK cells | From baseline throughout treatment period, up to 4 months
  Changes in Peripheral Blood Mononuclear Cells (PBMC) gene expression and flow cytometry patterns in NK cells.
Alterations of Avmacol® activity in PBMCs - T cells | From baseline throughout treatment period, up to 4 months
  Changes in Peripheral Blood Mononuclear Cells (PBMC) gene expression and flow cytometry patterns in T cells.
Change in serum cytokine levels | From baseline throughout treatment period, up to 4 months
  Change in serum cytokine levels, as determined by multiplexed bead-based cytokine assays.
Measurement of serum albumin-bound SF | From baseline throughout treatment period, up to 4 months
  Measurement of urinary metabolites of SF using isotope dilution mass spectrometry.
Safety profile in accordance with NCI CTCAE v.4 | Throughout treatment period, up to 4 months
  Patients will receive a diary for daily logging of adverse events. This will tabulated by Avmacol dose and type and grade of adverse events. The mean frequency and grade of events will be calculated by dose, and between-dose differences compared by means
Proportion of patients primary tumors harboring genomic alteration of NRF2 related genes | At baseline
  Genomic alterations in primary tumors will be characterized and the proportion determined by number of patients with NRF2 related genes per the total number of patients studied.

CONTACTS AND LOCATIONS:
Overall Officials: Dan P Zandberg, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - UPMC Eye Center - Eye and Ear Institute, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania